CLINICAL TRIAL: NCT06730334
Title: A Single Centre Prospective Cohort Study of Classification and Activity Assessment of Psoriatic Arthritis Based on Power Doppler (PD) Ultrasonography (PDUS)
Brief Title: Prospective Study of Classification and Activity Assessment of Psoriatic Arthritis Based on Power Doppler (PD) Ultrasonography (PDUS)
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Rui LIU, MD, MD, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2023-SR-415
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Psoriatic Arthritis; Secukinumab; Ultrasonography
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoriatic arthritis (PsA) is a complex inflammatory disease with heterogeneous clinical features, which complicates psoriasis in 30% of patients. PsA involves multiple tissues and clinical domains including skins and nails as well as arthritis, spondylitis, enthesitis, and dactylitis. Power Doppler (PD) ultrasonography (PDUS) is a sensitive non-invasive imaging technology used to assess disease activity and treatment response in PsA. This is a prospective, observational, open-label study to investigate disease activity, therapeutic response and bone destruction based on ultrasonography findings in patients with PsA.

ELIGIBILITY:
Inclusion Criteria:

* PsA patients as defined by CASPAR criteria
* Patients must be able to comply with the visit schedule, treatment plan, laboratory tests and other study procedures
* Patients must be given informed consent

Exclusion Criteria:

* History of other arthritis within the last 12 months
* Concomitant disease with acute or chronic infectious diseases
* Pregnancy or laction
* Poorly tolerated with venipuncture required for blood sampling during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult PsA patients as defined by CASPAR criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Madrid Sonographic Enthesitis Index (MASEI) | 12 weeks
  MASEI includes six entheses (the bilateral triceps, the quadriceps, both proximal and distal patellar and Achilles tendons and the proximal insertion of the plantar aponeurosis) and six elementary lesions (structure, thickening, erosion, enthesophytes, PD and bursa), with weighted punctuations that can be summed to a maximum score of 136.
DACTylitis glObal Sonographic (DACTOS) | 12 weeks
  DACTOS score will be used for every affected digit. There are four keys in DACTOS scoring: PTI（Peritendon extensor inflammation） evaluated in B-mode and PD at MCP and PIP joints level (maximum score, 4) STOe（Soft tissue oedema） evaluated in B-mode and PD in the most severely affected area of the digit (maximum score, 6) flexor tenosynovitis evaluated in B-mode and PD in the most severely affected area of the digit (maximum score, 6) EULAR-OMERACT combined score for synovitis evaluated at the MCP, PIP and DIP joints (maximum score, 9) DACTOS score summation ranges from 0 to 25 points. A DACTOS value<3 identified the US response.

SECONDARY OUTCOMES:
ACR20 Response | 12 weeks
  American College of Rheumatology (ACR) Response Criteria: An ACR20 response is defined as improvement of ≥20% from Baseline in the number of tender and swollen joints (from an analysis of 78 and 76 joints, respectively) and in three of the following five domains: a patient's global assessment of disease, a physician's global assessment of disease, and a patient's assessment of pain (all three measures evaluated on a visual-analogue scale of 0 to 100 mm), disability score on the Health Assessment Questionnaire-Disability Index (HAQ-DI; scores range from 0 to 3; higher scores indicate greater disability), and acute-phase reactants, as measured by high-sensitivity C-reactive protein (CRP) levels or erythrocyte sedimentation rate. An ACR50 response is defined as ≥50% improvement, and an ACR70 response is defined as ≥70% improvement in the above criteria.
Disease Activity Score 28-erythrocyte sedimentation rate (DAS28-ESR) | 12 weeks
  DAS28-ESR = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * GH. GH(mm)is general health using a visual analog scale (VAS) measuring general health (VAS-GH; 0 = best, 100 = worst)
Disease Activity Score 28-C-reactive protein (DAS28-CRP) | 12 weeks
  DAS28-CRP=0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28)+0.36×ln （CRP+1）+0.014* GH+0.96. GH(mm)is general health using a visual analog scale (VAS) measuring general health (VAS-GH; 0 = best, 100 = worst)
Disease Activity in PSoriatic Arthritis (DAPSA) | 12 weeks
  DAPSA score was calculated as the sum of: (1) SJC (range: 0-66), (2) TJC (range: 0-68), (3) patient pain assessment VAS measurement in centimeters (range: 0-10), (4) patient global assessment VAS measurement in centimeters (range: 0-10), and (5) serum acute-phase response, represented by CRP level in mg/dL (range: 0-10 mg/dL). The cut-off points for defining different disease activity are: ≤4, DAPSA-REM; >4 to ≤14, DAPSA-LDA; ≤14, DAPSA-REM+LDA; >14 to ≤28, DAPSA-MoDA; DAPSA-HAD, >28
ACR50 Response | 52 weeks
  American College of Rheumatology (ACR) Response Criteria: An ACR20 response is defined as improvement of ≥20% from Baseline in the number of tender and swollen joints (from an analysis of 78 and 76 joints, respectively) and in three of the following five domains: a patient's global assessment of disease, a physician's global assessment of disease, and a patient's assessment of pain (all three measures evaluated on a visual-analogue scale of 0 to 100 mm), disability score on the Health Assessment Questionnaire-Disability Index (HAQ-DI; scores range from 0 to 3; higher scores indicate greater disability), and acute-phase reactants, as measured by high-sensitivity C-reactive protein (CRP) levels or erythrocyte sedimentation rate. An ACR50 response is defined as ≥50% improvement, and an ACR70 response is defined as ≥70% improvement in the above criteria.
ACR70 Response | 52 weeks
  American College of Rheumatology (ACR) Response Criteria: An ACR20 response is defined as improvement of ≥20% from Baseline in the number of tender and swollen joints (from an analysis of 78 and 76 joints, respectively) and in three of the following five domains: a patient's global assessment of disease, a physician's global assessment of disease, and a patient's assessment of pain (all three measures evaluated on a visual-analogue scale of 0 to 100 mm), disability score on the Health Assessment Questionnaire-Disability Index (HAQ-DI; scores range from 0 to 3; higher scores indicate greater disability), and acute-phase reactants, as measured by high-sensitivity C-reactive protein (CRP) levels or erythrocyte sedimentation rate. An ACR50 response is defined as ≥50% improvement, and an ACR70 response is defined as ≥70% improvement in the above criteria.
Minimal disease activity (MDA) | 52 weeks
  MDA response was defined as achievement of at least five of the following seven criteria: TJC ≤1 (of 68), SJC ≤1 (of 66), PASI ≤1 or PsO affecting <3% BSA, patient pain VAS ≤15 mm, patient global disease activity VAS ≤20 mm, HAQ-DI ≤0.5, and tender entheseal points ≤1. Patients who met all seven MDA criteria were classified as achieving VLDA (very low disease activity)
Bone destruction | 52 weeks
  New bone destruction in x-ray, MRI, CT scan and ultrasonography. Based on New OMERACT definitions of US-detected pathologies, defined as intra- and/or extraarticular discontinuity of bone surface (visible in 2 perpendicular planes).
Bone destruction | 104 weeks
  New bone destruction in x-ray, MRI, CT scan and ultrasonography. Based on New OMERACT definitions of US-detected pathologies, defined as intra- and/or extraarticular discontinuity of bone surface (visible in 2 perpendicular planes).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Rheumatology and Immunology, Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu

REFERENCES:
- [Background] FitzGerald O, Ogdie A, Chandran V, Coates LC, Kavanaugh A, Tillett W, Leung YY, deWit M, Scher JU, Mease PJ. Psoriatic arthritis. Nat Rev Dis Primers. 2021 Aug 12;7(1):59. doi: 10.1038/s41572-021-00293-y. PMID 34385474
- [Background] Bruyn GA, Iagnocco A, Naredo E, Balint PV, Gutierrez M, Hammer HB, Collado P, Filippou G, Schmidt WA, Jousse-Joulin S, Mandl P, Conaghan PG, Wakefield RJ, Keen HI, Terslev L, D'Agostino MA; OMERACT Ultrasound Working Group. OMERACT Definitions for Ultrasonographic Pathologies and Elementary Lesions of Rheumatic Disorders 15 Years On. J Rheumatol. 2019 Oct;46(10):1388-1393. doi: 10.3899/jrheum.181095. Epub 2019 Feb 1. PMID 30709946
- [Background] Girolimetto N, Zabotti A, Tinazzi I, Possemato N, Costa L, Batticciotto A, Canzoni M, Citriniti G, De Lucia O, Figus F, Idolazzi L, McConnel R, Peluso R, Sakellariou G, Tullio A, Salvarani C, Scarpa R, Iagnocco A, Caso F, Macchioni P. Sensitivity to change and clinical correlations of the novel DACtylitis glObal Sonographic (DACTOS) score in psoriatic arthritis. Rheumatology (Oxford). 2021 Sep 1;60(9):4103-4111. doi: 10.1093/rheumatology/keaa885. PMID 33369655
- [Background] Zabotti A, Sakellariou G, Tinazzi I, Idolazzi L, Batticciotto A, Canzoni M, Carrara G, De Lucia O, Figus F, Girolimetto N, Macchioni P, McConnell R, Possemato N, Iagnocco A. Novel and reliable DACTylitis glObal Sonographic (DACTOS) score in psoriatic arthritis. Ann Rheum Dis. 2020 Aug;79(8):1037-1043. doi: 10.1136/annrheumdis-2020-217191. Epub 2020 May 19. PMID 32430315
- [Background] Coates LC, Nash P, Kvien TK, Gossec L, Mease PJ, Rasouliyan L, Pricop L, Jugl SM, Gandhi KK, Gaillez C, Smolen JS. Comparison of remission and low disease activity states with DAPSA, MDA and VLDA in a clinical trial setting in psoriatic arthritis patients: 2-year results from the FUTURE 2 study. Semin Arthritis Rheum. 2020 Aug;50(4):709-718. doi: 10.1016/j.semarthrit.2020.03.015. Epub 2020 May 15. PMID 32521325
- [Background] Mease P, van der Heijde D, Landewe R, Mpofu S, Rahman P, Tahir H, Singhal A, Boettcher E, Navarra S, Meiser K, Readie A, Pricop L, Abrams K. Secukinumab improves active psoriatic arthritis symptoms and inhibits radiographic progression: primary results from the randomised, double-blind, phase III FUTURE 5 study. Ann Rheum Dis. 2018 Jun;77(6):890-897. doi: 10.1136/annrheumdis-2017-212687. Epub 2018 Mar 17. PMID 29550766
- [Background] de Miguel E, Cobo T, Munoz-Fernandez S, Naredo E, Uson J, Acebes JC, Andreu JL, Martin-Mola E. Validity of enthesis ultrasound assessment in spondyloarthropathy. Ann Rheum Dis. 2009 Feb;68(2):169-74. doi: 10.1136/ard.2007.084251. Epub 2008 Apr 7. PMID 18390909
- [Background] Greenmyer JR, Stacy JM, Sahmoun AE, Beal JR, Diri E. DAS28-CRP Cutoffs for High Disease Activity and Remission Are Lower Than DAS28-ESR in Rheumatoid Arthritis. ACR Open Rheumatol. 2020 Sep;2(9):507-511. doi: 10.1002/acr2.11171. Epub 2020 Aug 29. PMID 32862564
- [Derived] Zhang Q, Mao C, Lu F, Wu Y, Ke Y, Liu R. Ultrasound dactylitis predicts bone erosion in early psoriatic arthritis: A longitudinal cohort study. Eur J Radiol. 2026 Jan 28;196:112704. doi: 10.1016/j.ejrad.2026.112704. Online ahead of print. PMID 41621380